CLINICAL TRIAL: NCT06720974
Title: AquaReBal - Aquatic Reactive Balance Training for Older Adults
Acronym: AquaReBal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Józef Piłsudski University of Physical Education (Other)
Collaborators: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Anna Ogonowska-Słodownik, Dr, Józef Piłsudski University of Physical Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-5483
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-12

CONDITIONS: Older Adults, Balance; Older People; Aquatic Physical Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AquaReBal - water-based RBT (Experimental): AquaReBal (water-based RBT) will be conducted at a warm therapy pool. Participants will not wear a safety harness in water as there is minimal risk of injury due to the water properties. The level of the water will be between umbilicus and xiphoid process to allow the participant to freely move in the standing position and ensure safety during perturbations. In addition, in the tasks that involve moving, the turbulence of the water will create additional perturbations.
  Interventions: Other: AquaReBal

INTERVENTIONS:
Other: AquaReBal — The interventions will be delivered one-on-one, in person at the KITE Research Institute by a trained and licensed physiotherapist. We will follow an RBT program previously developed by co-investigators. The interventions will be matched as closely as possible for frequency, intensity and time. The exercise interventions will be based on internal and external perturbations. Therapist-applied perturbations and multiple perturbation types and directions are of most benefit in terms of reactive balance control, so our study will focus on manual perturbations; the perturbations will be strong enough to cause stepping reactions. Interventions will be tailored to the individual participants' abilities.
  Each session will include a 10 min warm-up, at least 40 min of perturbations and a 10 min cool-down. Internal perturbations will be achieved by asking the participant to complete tasks that challenge balance control, such that they lose balance when attempting to perform the task.

SUMMARY:
Falls are the second leading cause of accidental injury deaths worldwide, mostly in older adults. Injuries resulting from a fall are a leading cause of hospitalizations among older adults in Canada with a higher total injury cost than any other cause of injury. People must often perform rapid and complex movements to keep from falling. Reactive balance training (RBT) is a type of training that focuses on improving an individual's ability to perform those types of movements and respond to unexpected or sudden changes. RBT and aquatic therapy were identified as a research priority for fall prevention. There is evidence that RBT reduces the rate of falls by a half in daily life and improvements in reactive balance are maintained up to a year after the end of the program. When RBT is conducted on land, some adverse events such as fear of falling and joint pain may occur. The water environment could minimize the limitations and barriers associated with land-based RBT. To date, there are no studies showing the effects of water-based RBT on reactive balance control in older adults.The study aims to explore if water-based RBT is a practical intervention to reduce the number of falls in older adults. Older adults will be recruited from the Greater Toronto Area. They will receive training 2 times per week for 6 weeks. The main practical factors around the intervention, such as how participants adhere to the treatment and how they accept the intervention will be measured. It will be assessed how the water-based and land-based RBT affects falls, balance, mobility and quality of life. With this study, the aim is to inform the way for a larger study targeting falls - one of the biggest problems among older adults.

DETAILED DESCRIPTION:
Background and Importance: Falls are the second leading cause of unintentional injury deaths worldwide, mostly in older adults. In 2018 falls in Canada had a higher total cost than any other cause of injury. Injuries resulting from a fall are a leading cause of hospitalizations among Canadian adults aged > 65 years. Recent clinical practice guidelines for older adults identified reactive balance training (RBT) and aquatic therapy as research priorities for fall prevention. There is evidence that RBT almost halves the rate of falls in daily life and improvements in reactive balance control are maintained even up to a year after the end of the program. When RBT is conducted on land, some adverse events (e.g. fear of falling and joint pain) occur. The water environment could minimize the limitations and barriers associated with land-based RBT. To date, there is a lack of studies reporting on the feasibility of conducting RBT in water for reactive balance control in older adults.

Goal(s) / Research Aims: Primary aim is to assess the feasibility AquaReBal intervention.

Methods / Approaches / Expertise: A single-arm pre-post study will be conducted among older adults. Participants will be recruited from the Greater Toronto Area. The intervention will be held twice per week for 6 weeks, 60 minutes per session. We will assess feasibility measures (indicators for process, resources, management, and safety parameters), reactive balance control and secondary outcome measures - history of falls, Physical Activity Scale for the Elderly (PASE), Activities-Specific Balance Confidence (ABC) Scale, European Quality of Life Instrument (EQ-5D), Mini Balance Evaluation Systems Test (mini-BESTest), Timed Up and Go (TUG) test. Participants' number of falls after intervention (6 weeks) until 6-month follow-up period will be monitored. Semi-structured interviews (qualitative component) will be conducted to understand the experiences of the participants with the interventions. Primary and secondary outcome measures will again be collected at 6 months post-intervention. The core research staff will consist of experts in the field of aquatic therapy and reactive balance. To facilitate knowledge translation after this study, we have adopted an integrated knowledge translation approach, including a patient partner and a knowledge user early in the preparation of this application and planning stages for the study.

Expected Outcomes: The proposed project will result in the development of a novel aquatic RBT. In addition, the participants' perspectives on the RBT training in water can provide further information on the feasibility of such interventions.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* able to stand ≥1 min
* able to independently walk ≥10 m without assistance
* a history of ≥2 falls in the past 12 months, history of an injurious fall in the past 12 months, and/or self-reported balance difficulties

Exclusion Criteria:

* Current diagnosis of neurological or sensory disorders
* uncorrected vision problems
* recurrent dizziness
* cognitive deficits
* medical conditions that could increase injury risk during balance tests (e.g. presence of a prior fragility fracture)
* conditions that would not allow the participant to get into the therapy pool (e.g. wounds, fear of water)
* currently attending physiotherapy or supervised exercise.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From enrollment to the end of treatment at 6 weeks and at 6 months post intervention
  Feasibility of recruitment, adherence and intervention fidelity will be measured. Because feasibility is a multidimensional construct we will also collect qualitative data about recruitment capability, randomization acceptability, data collection procedures and outcome measures, intervention delivery, intervention adherence and safety, barriers and facilitators to implementing the study, and retention of participants. Qualitative methods will include one-on-one interviews, unstructured observations, field notes and session recordings. We will use a flexible approach with regard to timing when qualitative data is collected as problems and implementation barriers arise; this will allow us to document information in real time, thus allowing us to make necessary refinements to the intervention and study protocol.

SECONDARY OUTCOMES:
Falls monitoring | From enrollment to the end of treatment at 6 weeks and 6 months post intervention
  The number of falls experienced by the participants will be monitored. Within 24 hours of experiencing a fall, the participants will complete a fall survey, either online or on paper. The survey will be composed of multiple-choice questions with closed-ended answers concerning the location of the fall and time of the day, as well as multiple-choice questions with an open-ended "other" option regarding the activity being performed at the time of the fall and potential contributing variables. In addition the survey will include questions about possible injuries from falling. A researcher will conduct monthly interviews with participants by phone or MS Teams to ensure the fall surveys are completed.
The Mini Balance Evaluation Systems Test (mini-BESTest) | From enrollment to the end of treatment at 6 weeks and 6 months post intervention
  The Mini Balance Evaluation Systems Test (mini-BESTest) is a 14-item observational rating scale that assesses systems underlying balance control, including reactive balance control and dynamic stability during walking. The Mini-BESTest is reliable and valid, and able to identify fall status in older people living in the community.
Timed Up and Go (TUG) | From enrollment to the end of treatment at 6 weeks and at 6 months post intervention
  Timed Up and Go (TUG) is a commonly-used screening tool for fall risk in the inpatient and community setting. A faster time indicates better functional performance and a score of ≥13.5 s is used as a cut-point to identify those at increased risk of falls. The TUG test has shown acceptable psychometric properties and is considered appropriate for the general older adult population.
Physical activity | From enrollment to the end of treatment at 6 weeks and at 6 months post intervention
  The Physical Activity Scale for the Elderly (PASE) is a 12-item reliable and valid self-report instrument specifically designed for older adults. It is used to assess physical activity over a one-week time period.
Psychological consequences | From enrollment to the end of treatment at 6 weeks and 6 months post intervention
  The Activities-Specific Balance Confidence scale (ABC scale) is a self-report measure where participants rate their confidence in performing daily tasks while standing and walking using percentages, with higher percentages indicating more confidence. The ABC scale demonstrated strong internal consistency reliability in community-dwelling older adults.
Health-related quality of life | From enrollment to the end of treatment at 6 weeks and 6 months post intervention
  5-level EuroQoL is simple measure of health-related quality of life and has been used widely in older adults.
Reactive balance control | From enrollment to the end of treatment at 6 weeks and 6 months post intervention
  To assess reactive balance control, participants will be outfitted with reflective markers and complete 8-10 walking trials on a movable platform. In two trials, the platform will move forward suddenly on heel strike to trigger a slip-like perturbation. In two other trials, the platform will move backward suddenly on toe-off to trigger a trip-like perturbation. The perturbation waveform will consist of a 300 ms square-wave acceleration, followed immediately by 300 ms deceleration. The remaining four to six trials will consist of unperturbed walking. The slip/trip and unperturbed walking trials will be presented in pseudorandom order. Reactive balance will be measured using three-dimensional motion capture (Vicon Motion Systems, Oxford, UK), and force plates (AMTI, Watertown, MA, USA). When responding to the perturbation, biomechanical stability will be measured using an established method that considers the distance between the center of mass and base of support.

IPD SHARING:
Plan to Share IPD: Undecided